CLINICAL TRIAL: NCT02989415
Title: Assessment of Ventilatory Management During General Anesthesia for Robotic Surgery and Its Effects on Postoperative Pulmonary Complications: A Prospective Observational Multicenter Study
Brief Title: Assessment of Ventilatory Management During General Anesthesia for Robotic Surgery
Acronym: AVATaR
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Genova (Other); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Ary Serpa Neto, MD, MSc, PhD, Hospital Israelita Albert Einstein
Other Study IDs: AVATaR
Record Dates: First submitted 2016-12-07; First posted 2016-12-12 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Robotic Surgery; Mechanical Ventilation
Keywords: Anesthesia; Mechanical Ventilation; Robotic Surgery; Postoperative Pulmonary Complications
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanical Ventilation: Patients undergoing mechanical ventilation during robotic surgery
  Interventions: Other: Mechanical Ventilation

INTERVENTIONS:
Other: Mechanical Ventilation — Mechanical ventilation during robotic surgery

SUMMARY:
The aim of this study is to assess the incidence of postoperative pulmonary complications in patients undergoing mechanical ventilation during general anesthesia for robotic surgery, to characterize current practices of mechanical ventilation and to evaluate a possible association between ventilatory parameters and postoperative pulmonary complications.

DETAILED DESCRIPTION:
Research questions:

1. What is the incidence of PPC in patients undergoing mechanical ventilation during general anesthesia for robotic surgery?
2. Are the outcomes in patients undergoing robotic surgery dependent on ventilation practice and surgical positioning?
3. What is the incidence of patients at high risk for PPC undergoing robotic surgery

Methods:

In this international observational study, consecutive patients undergoing mechanical ventilation for robotic surgery are eligible for participation. Patients in participating centers will be screened on a daily basis. Patients undergoing mechanical ventilation for robotic surgery will be included during a 30-day period. The inclusion period will be flexible for participating centers and determined at a later stage together with the study-coordinator.

Time points of data collection:

1. Demographic data and baseline data, including severity scores (e.g. ASA) and ARISCAT, are collected from the clinical files on the day of surgery
2. Ventilation settings, gas exchange variables, positioning and vital parameters are collected hourly during surgery
3. Chest radiography data from available chest X-rays (i.e., no extra chest X-rays are obtained)
4. Predefined complications are recorded from medical chart until the first five postoperative days, discharge from hospital or death, whatever comes first
5. Length of hospital stay, and hospital mortality

Centres: The investigators aim to recruit 20 - 50 centers worldwide.

Ethics Approval: National coordinators will be responsible for clarifying the need for ethics approval and applying for this where appropriate according to local policy. Centres will not be permitted to record data unless ethics approval or an equivalent waiver is in place. The investigators expect that in most, if not every participating country, a patient informed consent is not be required.

Monitoring: Due to the observational nature of the study, a DSMB is not be necessary.

Study Population: Adult patients undergoing mechanical ventilation for robotic surgery.

Data Collection: Data will be collected at inclusion, during surgery and every day during five days, and day of hospital discharge. Data will be coded by a patient identification number (PIN) of which the code will be kept safe at the local sites. The data will be transcribed by local investigators onto an internet based electronic CRF.

Sample Size Calculation: A formal sample size will not be calculated, seen the largely descriptive character of this investigation. Data from 500 patients is expected to be collected, which will be sufficient to test the hypotheses.

Statistical Analysis: Patient characteristics will be compared and described by appropriate statistics. Student's t-test or Mann-Whitney U-tests are used to compare continuous variables and chi-squared tests are used for categorical variables. Data are expressed as means (SD), medians (interquartile range) and proportions as appropriate. Comparisons between and within groups are performed using one-way ANOVA and post-hoc analyses for continuous variables.

The primary analysis concerns the determination of the incidence of postoperative pulmonary complications in patients undergoing mechanical ventilation for robotic surgery.

To identify potential factors associated with outcome like development of postoperative pulmonary complications, or death, univariable analyses will be performed. A multi-level multivariable logistic regression model will be used to identify independent risk factors. A gradual approach will be used to enter new terms into the model, with a limit of p < 0.2 to enter the terms. Time to event variables will be analyzed using Cox regression and visualized by Kaplan-Meier.

Organization: The study is conducted by the PROtective VEntilation Network (PROVENet). National co-ordinators will lead the project within individual nations and identify participating hospitals, translate study paperwork, distribute study paperwork and ensure necessary regulatory approvals are in place. They provide assistance to the participating clinical sites in trial management, record keeping and data management. Local coordinators in each site will supervise data collection and ensure adherence to Good Clinical Practice during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* All surgical procedures performed under general anesthesia for robotic surgery, including head and neck operations, chest, cardiac, and abdominal surgeries

Exclusion Criteria:

* Any procedure during pregnancy
* Procedures outside of the operating room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing mechanical ventilation during general anesthesia for robotic surgery
Sampling Method: Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications | Five days or until hospital discharge, whichever occurs first
  Composite of five postoperative pulmonary complications

SECONDARY OUTCOMES:
Mechanical ventilation practice | Intraoperatively
  Mechanical ventilation practice in patients submitted to general anesthesia for robotic surgery
Mechanical ventilation practice and postoperative pulmonary complications | Five days or until hospital discharge, whichever occurs first
  Association between mechanical ventilation practice and development of postoperative pulmonary complications
Surgical positioning and ventilation | Intraoperatively
  Association between surgical positioning and ventilatory parameters
Patients at high risk for postoperative pulmonary complications | Pre-operatively
  Incidence of patients at high risk for postoperative pulmonary complications according to the ARISCAT score
Mechanical ventilation practice and intraoperative complications | Intraoperatively
  Association between mechanical ventilation practice and development of intraoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Ary Serpa Neto, MD, MSc, PhD, Study Chair — Department of Critical Care Medicine, Hospital Israelita Albert Einstein; Veronica NF Queiroz, MD, Study Director — AVATaR Study Coordinator, Anesthesiology, Hospital Israelita Albert Einstein; Luiz Guilherme V da Costa, MD, PhD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; Rogério P Barbosa, MD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; Flavio Takaoka, MD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; Luc de Baerdemaeker, MD, PhD, Principal Investigator — Department of Anesthesiology and Perioperative Medicine; Ghent University Hospital - Ghent University; Ghent, Belgium; Daniel S Cesar, MD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; Ulisses C D'Orto, MD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; José Roberto Galdi, MD, PhD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; Vijaya Gottumukkala, MD, PhD, Principal Investigator — Department of Anesthesiology and Perioperative Medicine; The University of Texas MD Anderson Cancer Center; Houston, Texas, USA; Sabrine NT Hemmes, MD, PhD, Principal Investigator — Department of Anaesthesiology; Academic Medical Center; University of Amsterdam; Amsterdam, The Netherlands; Markus W Hollmann, MD, PhD, Principal Investigator — Department of Anaesthesiology; Academic Medical Center; University of Amsterdam; Amsterdam, The Netherlands; Alain Kalmar, MD, PhD, Principal Investigator — Department of Anesthesia and Intensive Care Medicine; Maria Middelares Hospital; Ghent, Belgium; Renato M Mariano, MD, PhD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; Idit Matot, MD, PhD, Principal Investigator — Division of Anesthesiology, Intensive Care and Pain; Tel Aviv Medical Center and the Sackler Faculty of Medicine; Tel Aviv University; Tel Aviv, Israel; Guido Mazzinari, MD, Principal Investigator — Department of Anaesthesiology; Manises General Hospital; Manises, Spain; Gary H Mills, MD, PhD, Principal Investigator — Department of Anaesthesia and Critical Care Medicine; Sheffield Teaching Hospital; Sheffield, UK; Irimar P Posso, MD, PhD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; Alexandre Teruya, MD, PhD, Principal Investigator — Anesthesiology, Hospital Israelita Albert Einstein; Marcos Francisco Vidal Melo, MD, PhD, Principal Investigator — Department of Anesthesia, Critical Care and Pain Medicine; Massachusetts General Hospital; Harvard Medical School; Boston, MA, USA; Paolo Pelosi, MD, FERS, Principal Investigator — Department of Surgical Sciences and Integrated Diagnostics; IRCCS San Martino IST; University of Genoa; Genoa, Italy; Marcelo Gama de Abreu, MD, PhD, Principal Investigator — Pulmonary Engineering Group; Department of Anesthesiology and Intensive Care Medicine; University Hospital Carl Gustav Carus; Technische Universität Dresden; Dresden, Germany; Marcus J Schultz, MD, PhD, Principal Investigator — Department of Intensive Care; Academic Medical Center; University of Amsterdam; Amsterdam. The Netherlands
Locations (12):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Maria Middelares Hospital, Ghent, Belgium
- Hospital Israelita Albert Einstein, São Paulo, Brazil
- Germany (2):
  - University of Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Essen
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Spain (2):
  - Hospital Clinico Universitario San Carlos, Madrid, Madrid
  - Hospital Clinic of Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
The data will be available for substudies suggested by members of the collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the publication of the main manuscript
Access Criteria: The data will be available for substudies suggested by members of the collaboration.

REFERENCES:
- [Result] Neto AS, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Gajic O, El-Tahan MR, Ghamdi AA, Gunay E, Jaber S, Kokulu S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Ranieri VM, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Amato MB, Costa EL, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Association between driving pressure and development of postoperative pulmonary complications in patients undergoing mechanical ventilation for general anaesthesia: a meta-analysis of individual patient data. Lancet Respir Med. 2016 Apr;4(4):272-80. doi: 10.1016/S2213-2600(16)00057-6. Epub 2016 Mar 4. PMID 26947624
- [Result] Serpa Neto A, Schultz MJ, Gama de Abreu M. Intraoperative ventilation strategies to prevent postoperative pulmonary complications: Systematic review, meta-analysis, and trial sequential analysis. Best Pract Res Clin Anaesthesiol. 2015 Sep;29(3):331-40. doi: 10.1016/j.bpa.2015.09.002. Epub 2015 Sep 18. PMID 26643098
- [Result] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Biehl M, Binnekade JM, Canet J, Fernandez-Bustamante A, Futier E, Gajic O, Hedenstierna G, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Putensen C, Ranieri M, Scavonetto F, Schilling T, Schmid W, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network Investigators. Protective versus Conventional Ventilation for Surgery: A Systematic Review and Individual Patient Data Meta-analysis. Anesthesiology. 2015 Jul;123(1):66-78. doi: 10.1097/ALN.0000000000000706. PMID 25978326
- [Result] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Moine P, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network investigators. Incidence of mortality and morbidity related to postoperative lung injury in patients who have undergone abdominal or thoracic surgery: a systematic review and meta-analysis. Lancet Respir Med. 2014 Dec;2(12):1007-15. doi: 10.1016/S2213-2600(14)70228-0. Epub 2014 Nov 13. PMID 25466352
- [Result] Hemmes SN, Serpa Neto A, Schultz MJ. Intraoperative ventilatory strategies to prevent postoperative pulmonary complications: a meta-analysis. Curr Opin Anaesthesiol. 2013 Apr;26(2):126-33. doi: 10.1097/ACO.0b013e32835e1242. PMID 23385321
- [Result] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Result] Danic MJ, Chow M, Alexander G, Bhandari A, Menon M, Brown M. Anesthesia considerations for robotic-assisted laparoscopic prostatectomy: a review of 1,500 cases. J Robot Surg. 2007;1(2):119-23. doi: 10.1007/s11701-007-0024-z. Epub 2007 May 30. PMID 25484947
- [Result] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Result] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Derived] Serafini SC, Hemmes SNT, Serpa Neto A, Schultz MJ, Tschernko E, Gama de Abreu M, Mazzinari G, Ball L; LAS VEGAS - and the AVATaR - investigators. Risk factors for PPCs in laparoscopic non-robotic vs. laparoscopic robotic abdominal surgery (LapRas): rationale and protocol for a patient-level analysis of LAS VEGAS and AVATaR. Rev Esp Anestesiol Reanim (Engl Ed). 2024 Oct;71(8):592-600. doi: 10.1016/j.redare.2024.07.001. Epub 2024 Jul 8. PMID 38987020
- [Derived] Assessment of Ventilation during general AnesThesia for Robotic surgery (AVATaR) Study Investigators; PROtective VEntilation (PROVE) Network; Writing Committee Members; Steering Committee Members; AVATaR Investigators. Ventilation and outcomes following robotic-assisted abdominal surgery: an international, multicentre observational study. Br J Anaesth. 2021 Feb;126(2):533-543. doi: 10.1016/j.bja.2020.08.058. Epub 2020 Oct 31. PMID 33131757
- [Derived] Queiroz VNF, da Costa LGV, Barbosa RP, Takaoka F, De Baerdemaeker L, Cesar DS, D'Orto UC, Galdi JR, Gottumukkala V, Cata JP, Hemmes SNT, Hollman MW, Kalmar A, Moura LAB, Mariano RM, Matot I, Mazzinari G, Mills GH, Posso IP, Teruya A, Vidal Melo MF, Sprung J, Weingarten TN, Treschan TA, Koopman S, Eidelman L, Chen LL, Lee JW, Arino Irujo JJ, Tena B, Groeben H, Pelosi P, de Abreu MG, Schultz MJ, Serpa Neto A; AVATaR and PROVE Network investigators. International multicenter observational study on assessment of ventilatory management during general anaesthesia for robotic surgery and its effects on postoperative pulmonary complication (AVATaR): study protocol and statistical analysis plan. BMJ Open. 2018 Aug 23;8(8):e021643. doi: 10.1136/bmjopen-2018-021643. PMID 30139899
- See also: Hospital Israelita Albert Einstein — http://www.einstein.br

DOCUMENTS (2):
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT02989415/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT02989415/SAP_001.pdf